CLINICAL TRIAL: NCT06689865
Title: Effectiveness Trial to Examine the Emerging Service Delivery Models for Over-the-Counter (OTC) Hearing Aids
Brief Title: Innovations in Hearing Accessibility and Technology (IHAT) Study
Acronym: IHAT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-2351; R01DC021653 (NIH)
Record Dates: First submitted 2024-11-13; First posted 2024-11-15 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Hearing Loss; Hearing Aids; OTC Hearing Aids
Keywords: hearing loss; hearing aids; OTC hearing aids; service delivery models; effectiveness trial; Over-the-counter hearing aids
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- HA-HCP (Active Comparator)
  Interventions: Device: HA-HCP
- OTC-HCP (Experimental)
  Interventions: Device: OTC-HCP
- OTC-R (Experimental)
  Interventions: Device: OTC-R
- OTC-SF (Active Comparator)
  Interventions: Device: OTC-SF

INTERVENTIONS:
Device: HA-HCP — Prescription hearing aid fit by a hearing healthcare professional using audiology best practices.
  Arms: HA-HCP
Device: OTC-HCP — Over-the-counter hearing aids fit by a hearing care professional using audiology best practices.
  Arms: OTC-HCP
Device: OTC-R — OTC fit to an individual using some best practices via remote consultation.
  Arms: OTC-R
Device: OTC-SF — Self-fit OTC hearing aids without any clinical support from HCPs.
  Arms: OTC-SF

SUMMARY:
The research will explore outcomes of different service delivery models of over-the-counter (OTC) hearing aids by comparing them to prescription hearing aids fitted by specialists in individuals with mild to moderate hearing loss. The investigators will examine how each type affects users' experiences, behavior, thinking skills, and brain activity related to hearing. Additionally, the study will focus on what types of people prefer each hearing aid option, what helps or hinders these choices, and compare the costs of four different service options. This approach will help transition from research findings into real-world practice, providing useful information for healthcare providers and policymakers about OTC hearing aid options.

DETAILED DESCRIPTION:
The aim of the proposed project is to evaluate the effectiveness of emerging over-the-counter (OTC) service delivery models with the gold standard traditional prescription hearing aids fit by hearing care professionals (HCP) using audiology best practices. OTC service delivery models include OTC HA fit to individual users using best practices with in person HCP support (OTC-HPC), via remote consultation (OTC-R) and self-fit OTC HAs without any clinical support (OTC-SF). The study will use a prospective four-arm randomized controlled trial design with longitudinal repeated measures.

ELIGIBILITY:
Inclusion Criteria:

* Adult onset, bilateral, mild-to-moderate sensorineural hearing loss documented by audiological evaluation
* Aged 40 years or older
* No previous HA experience greater than 3 months
* Able to read and understand patient education materials
* Willing to be randomized to one of the four groups, and
* Owns a smartphone

Exclusion Criteria:

* Hearing loss that is too severe for OTC HAs
* Middle ear disorders or conductive pathology present
* Asymmetrical hearing loss
* Diagnosed neurological condition such as dementia or Parkinson's disease or a score lower than 25 on the MOCA
* Non-English speaking as it may impact the ability to complete our test battery

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2024-11-13 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Abbreviated Profile of Hearing Aid Benefit (APHAB) | T0 = Baseline, T1 = 6 months post intervention, T2 = 12 months post intervention
  It is a 24-item self-reported measure of hearing disability and hearing aid benefit. It includes four subscales that address different listening challenges: ease of communication, reverberation, background noise, and aversiveness of sounds, with each subscales comprising six items. The ease of communication, reverberation, and background noise primarily measure challenges related to speech communication. The global score on the APHAB is the average of these three subscale scores. The hearing aid benefit is calculated by comparing the difficulty level reported without amplification (unaided) to the difficulty level with amplification (aided). Scores range from 1% to 99%, with higher scores indicating greater perceived hearing difficulty.

SECONDARY OUTCOMES:
Satisfaction with Amplification in Daily Living (SADL) | T0= Baseline, T1= 6 months post intervention, T2= 12 months post intervention
  SADL is a 15-item self-reported outcome measure that evaluates an individual's satisfaction with their hearing aids on a 7-point rating scale. The questionnaire is divided into four subscales. The positive effect subscale quantifies improved performance with hearing aids. The personal image subscale quantifies self-image and stigma. The negative feature subscale evaluates undesirable aspects of using hearing aids. The service and cost subscale assesses the adequacy of the professional's service and the device's cost. Higher scores indicate greater satisfaction with hearing aids.
Revised Hearing Handicap Inventory -Screening (RHHI-S) | T0= Baseline, T1= 6 months post intervention, T2= 12 months post intervention
  It is a 10-item self-perceived hearing handicap measure that can be used for adults of all ages. The response options on this scale are yes (4), sometimes (2), and no (0), and ranges from 0 to 40. The total score is the sum of all the responses, with higher scales indicating greater perceived difficulties.
Patient Global Impression of Change (PGI-C) | T1= 6 months post intervention, T2= 12 months post intervention
  PGI-C assesses the patient's belief about the efficacy of treatment with a single-item questionnaire on a 7-point rating scale. Lower scores indicate improved outcomes.
Connected Speech Test (CST) | T0= Baseline, T1= 6 months post intervention, T2= 12 months post intervention
  The connected speech test is a sentence intelligibility test consisting of 48 passages with 8-10 sentences of a connected discourse spoken by a female speaker. A pair of passages will be presented to the participant, and the 25 keywords in each passage will be scored for percentage correct score. A higher percentage correct score indicates higher sentence intelligibility.
Quick Speech in Noise (QuickSIN) | T0= Baseline, T1= 6 months post intervention, T2= 12 months post intervention
  It assesses the patient's ability to hear in background noise. The patient repeats sentences that are embedded in different noisy environments and the result is a signal-to-noise ratio loss. The test stimuli are pre-recorded sentences embedded in speech babble at varying signal-to-noise ratios from easy to very difficult.

CONTACTS AND LOCATIONS:
Overall Officials: Vinaya Manchaiah, AuD, MBA, PhD, Principal Investigator — University of Colorado, Denver; Anu Sharma, PhD, Principal Investigator — University of Colorado, Boulder
Locations (2):
- United States (2):
  - University of Colorado School of Medicine, Aurora, Colorado
  - University of Colorado Boulder, Boulder, Colorado

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Background] De Sousa KC, Manchaiah V, Moore DR, Graham MA, Swanepoel W. Effectiveness of an Over-the-Counter Self-fitting Hearing Aid Compared With an Audiologist-Fitted Hearing Aid: A Randomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2023 Jun 1;149(6):522-530. doi: 10.1001/jamaoto.2023.0376. PMID 37052929
- [Background] De Sousa KC, Manchaiah V, Moore DR, Graham MA, Swanepoel W. Long-Term Outcomes of Self-Fit vs Audiologist-Fit Hearing Aids. JAMA Otolaryngol Head Neck Surg. 2024 Sep 1;150(9):765-771. doi: 10.1001/jamaoto.2024.1825. PMID 38990557
- [Background] Knoetze M, Manchaiah V, De Sousa K, Moore DR, Swanepoel W. Comparing Self-Fitting Strategies for Over-the-Counter Hearing Aids: A Crossover Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2024 Sep 1;150(9):784-791. doi: 10.1001/jamaoto.2024.2007. PMID 39052241